CLINICAL TRIAL: NCT06924151
Title: the Prospective, Randomized, Controlled, Multi-center Study to Establish the Safety and Effectiveness of Isolated Surgical Aortic Valve Replacement in Low Risk Patients Who Have Symptomatic Severe Aortic Stenosis
Brief Title: Isolated Surgical Aortic Valve Replacement in Low Risk AS Patients
Acronym: AMETHYST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMETHYST-001
Record Dates: First submitted 2025-02-11; First posted 2025-04-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical aortic valve replacement (Experimental): Surgical aortic valve replacement (SAVR) with free choice of surgical bioprosthesis and free choice of surgical access according to the surgeon's preference
  Interventions: Procedure: surgical aortic valve replacement
- Transcatheter aortic valve replacement (Active Comparator): Transcatheter aortic valve replacement (TAVR) using the device available in Japan in facilities approved to perform TAVR.
  Interventions: Procedure: Transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: surgical aortic valve replacement — SAVR
  Arms: Surgical aortic valve replacement
Procedure: Transcatheter aortic valve replacement — TAVR
  Arms: Transcatheter aortic valve replacement

SUMMARY:
To establish the safety and effectiveness of surgical aortic valve replacement (SAVR) in patients with isolated severe, calcific aortic stenosis who are at low surgical risk.

DETAILED DESCRIPTION:
This study is the Prospective, Randomized, Controlled, Multi-center Study of Isolated SAVR in Low Risk AS Patients (The AMETHYST trial). Patients will be randomized 1:1 to receive either SAVR or transcatheter heart valve replacement (TAVR) with a commercially available surgical and transcatheter bioprosthetic valves. The aim of this study was to assess the non-inferiority of SAVR compared with TAVR for the combined endpoints of death from any cause, stroke and rehospitalization (hospitalization related to biological valves or procedures or heart failure) at 1 year postoperatively. Patients will be seen for follow-up visits at discharge, 30 days, and annually through 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. All study participants must meet the following inclusion criteria 1. Severe, calcific aortic stenosis with the following criteria:

   * Jet velocity ≥4.0 m/s or mean gradient ≥ 40 mmHg OR
   * AVA ≤1.0 cm2 or AVA index ≤ 0.6 cm2/m2 Note: Qualifying TTE must be within 90 days prior to randomization

   AND 2. NYHA class ≥ II OR Exercisee test that demonstrates a limited exercise capacity, abnormal blood pressure response, or arrhythmia OR Asymptomatic patients with LVEF <50%
2. The Heart Team agrees that the surgical mortality risk is less than 4% according to STS-PROM. The Heart Team's assessment should include evaluation of overall clinical status and comorbidities that may not be adequately captured by risk calculators such as STS-PROM, in addition to the risk score itself.
3. The patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by certified review board.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

1. History of cardiovascular surgery or thoracotomy
2. Pre-existing other valvular disease, coronary artery disease or aortic disease required intervention Note: interventions for arrhythmia or root enlargement are not considered exclusionary.
3. Heart Team assessment that chest abnormalities or significant frailty would prevent safe SAVR.
4. Native aortic annulus size unsuitable for sizes the currently approved and marketed SAVR or TAVR based on preoperative 3D-CT image analysis.
5. Iliofemoral vessel characteristics that whould preclude safe insertion of the introducer sheath.
6. Evidence of an acute myocardial infarction or PCI ≤ 30 days before randomization
7. Aortic valve is unicuspid
8. Severe aortic regurgitation (>3+)
9. Severe mitral regurgitation (>3+) or ≥ moderate stenosis
10. Severe tricuspid regurgitation (>3+) or ≥ moderate stenosis
11. Pre-existing mechanical or bioprosthetic valve in any position.
12. Complex coronary artery disease:

    1. Heart Team assessment that CABG is recommended at the time of SAVR
    2. Heart Team assessment that optimal revascularization cannot be performed
13. Symptomatic carotid or vertebral artery disease or treatment of carotid stenosis within 30 days of randomization
14. Leukopenia (WBC < 3000 cell/mL), Thrombocytopenia (Plt < 50,000 cell/mL), history of bleeding diathesis or coagulopathy.
15. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of randomization
16. Hypertrophic cardiomyopathy with obstruction (HOCM)
17. Ventricular dysfunction with LVEF < 30%
18. Cardiac imaging (echo, CT, and/or MRI) evidence of intracardiac mass, thrombus or vegetation
19. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure
20. Stroke or transient ischemic attack (TIA) within 90 days of randomization
21. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy
22. Active bacterial endocarditis within 180 days of randomization
23. Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen
24. Severe pulmonary hypertension (e.g., PA systolic pressure ≥ 2/3 systemic pressure)
25. History of cirrhosis or active liver disease
26. Significant abdominal or thoracic aortic disease (such as porcelain aorta, aneurysm, severe calcification, aortic coarctation, etc.) that would preclude cannulation and aortotomy for SAVR or safe passage of the delivery system for TAVR.
27. Patient refuses blood products.
28. BMI > 50 kg/m2
29. Estimated life expectancy < 24 months.
30. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication.
31. Immobility or significant cognitive impairment that would prevent completion of study procedure.
32. Currently participating in an investigational drug or another device study.
33. Unsuitable as candidates by the principal investigator or a research associate for other reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2037-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause mortality, all stroke, and rehospitalization (valve-related or procedure-related and including heart failure) | at 1 year post procedure

SECONDARY OUTCOMES:
the rate of all-cause mortality or disabling stroke | at one year
the rate of all-cause mortality | at one year
the rate of all stroke | at one year
the rate of disabling stroke | at one year
the rate of rehospitalization (valve-related or procedure-related and including heart failure) | at one year
the rate of new bundle branch block or new pacemaker implantation | at one year
the rate of new onset of atrial fibrillation | at 30 days
the rate of life-threatening bleeding | at one year
the rate of occurrence of perivalvular regurgitation ≥ mild by echocardiography | at one year
Quality of life as assessed by KCCQ | at one year
Quality of life as assessed by EQ-5D-5L | at one year
the rate of prosthetic valve endocarditis | at one year
the rate of prosthetic valve thrombosis | at one year
the rate of valve-related dysfunction requiring repeat procedure | at one year

OTHER OUTCOMES:
All cause mortality | at 30 days
The rate of all stroke (disabling and nondisabling) | at 30 days
The rate of Rehospitalization (valve-related or procedure-related and including heart failure) | at 30 days
All cause mortality or all stroke | at one year
All cause mortality or disabling stroke | at 30 days
The rate of vascular complications (major) | at 30 days and one year
The rate of Bleeding complications (life threatening, disabling or major) | at 30 days
The rate of myocardial infarction | at 30 days and one year
The rate of acute kidney injury | at 30 days
the rate of new bundle branch block or new pacemaker implantation | at 30 days
the rate of occurrence of perivalvular regurgitation ≥ mild by echocardiography | at 30 days
The rate of coronary obstruction requiring intervention | at 30 days and one year
New York Heart Association class | at 30 days and one year
  NYHA Classification criteria:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity Class II: Subjects with cardiac disease resulting in slight limitation of physical activity Class III: Subjects with cardiac disease resulting in marked limitation of physical activity Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort
Six-minute walk test | at 30 days and one year
The length of postoperative ICU stay | up to one year
Discharge location | up to one year
  * Home [including return to pre-admission facilities (excluding hospitals)]
  * Other hospital [excluding rehabilitation hospital]
  * Rehabilitation hospital
  * Death
  * Other
Health status as evaluated by Quality of Life questionnaires (KCCQ) | at 30 days
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.
  This instrument was developed and validated by John Spertus. John is Director of Cardiovascular Education and Outcomes Research at the Mid America Heart Institute, and he is also a Professor of Medicine at the University of Missouri - Kansas City.
  In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. For brevity, only the performance characteristics of the overall summary score are presented in this discussion.
Health status as evaluated by Quality of Life questionnaires (EQ-5D-5L) | at 30 days
  EQ-5D-5L: Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state
Cognitive function assessed by the MMSE | at one year
  It is an 11-question measure that tests five areas of cognitive function:
  orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
The rate of new onset atrial fibrillation | at one year
Endpoints of minimally invasive aortic valve replacement (MICS AVR) vs TAVR | at 30 days and one year

CONTACTS AND LOCATIONS:
Locations (37):
- Japan (37):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - New Tokyo Hospital, Matsudo, Chiba
  - Chibanishi General Hospital, Matsudo, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Fukui Cardiovascular center, Fukui-shi, Fukui
  - Kyushu Univerisity, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Kurume University, Kurume, Fukuoka
  - Hyogo Medical University, Nishinomiya, Hyōgo
  - Kagoshima Medical Center, Kagoshima, Kagoshima-ken
  - Tokai University, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kawasakisaiwai Hospital, Kawasaki, Kanagawa
  - St.Marianna University School of Medicine, Kawasaki, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Kumamoto University, Kumamoto, Kumamoto
  - Shinshu University, Matsumoto, Nagano
  - Nagasaki University, Nagasaki, Nagasaki
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Yuuai Medical Center, Tomigusuku, Okinawa
  - Kishiwada Tokusyukai Hospital, Kishiwada, Osaka
  - Osaka International Medical and Science Center, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Kinki University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University Shool of Medicine, Hamamatsu, Shizuoka
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical University, Shimotsuga, Tochigi
  - Tokushima University, Tokushima, Tokushima
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Tokyo Women's Medical University, Shinjuku, Tokyo
  - Tottori University, Yonago, Tottori
  - Wakayama Medical University, Wakayama, Wakayama
  - Oita University, Ōita, Yufu

IPD SHARING:
Plan to Share IPD: No